CLINICAL TRIAL: NCT03840200
Title: A Phase Ib, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Ipatasertib in Combination With Rucaparib in Patients With Advanced Breast, Ovarian, or Prostate Cancer
Brief Title: A Study Evaluating the Safety, Pharmacokinetics and Efficacy of Ipatasertib Administered in Combination With Rucaparib in Participants With Advanced Breast, Ovarian Cancer, and Prostate Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BO40933
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Prostate Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms | interventions — ipatasertib; rucaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose escalation-Cohort 1 (Experimental): Participants with advanced breast cancer, ovarian cancer, or prostate cancer will receive ipatasertib, 300 milligrams (mg), orally, once daily (QD) for 7 days in the run-in period. Participants will then receive ipatasertib, 300 mg, orally QD, and rucaparib, 400 mg, orally twice daily (BID) in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Rucaparib
- Dose escalation-Cohort 2a (Experimental): Participants with advanced breast cancer, ovarian cancer, or prostate cancer will receive ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants will then receive ipatasertib, 300 mg, orally QD, and rucaparib, 600 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Rucaparib
- Dose escalation-Cohort 2b (Experimental): Participants with advanced breast cancer, ovarian cancer, or prostate cancer will receive ipatasertib, 400 mg, orally, QD for 7 days in the run-in period. Participants will then receive ipatasertib, 400 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Rucaparib
- Dose escalation-Cohort 3 (Experimental): Participants with advanced breast cancer, ovarian cancer, or prostate cancer are planned to receive ipatasertib 400 mg orally QD for 7 days (run-in period prior to Cycle 1). Participants will then receive ipatasertib 400 mg orally QD and rucaparib 600 mg, orally BID in 28 days cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Rucaparib
- Dose Expansion (Experimental): The recommended dose (ipatasertib and rucaparib) identified in Part 1 will be evaluated in participants with advanced prostate cancer who have had at least one line of prior therapy with second-generation androgen-receptor (AR)-targeted agents (e.g., abiraterone, enzalutamide, apalutamide).
  Interventions: Drug: Ipatasertib; Drug: Rucaparib

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered orally.
  Other Names: RO5532961, GDC-0068
Drug: Rucaparib — Rucaparib will be administered orally.
  Other Names: CO-338

SUMMARY:
This is a study in participants with advanced breast, ovarian, or prostate cancer to investigate the dose, safety, pharmacokinetics, and preliminary efficacy of ipatasertib in combination with rucaparib. The study consists of two parts: a Dose-Escalation Phase (Part 1) in participants with previously treated advanced breast cancer, ovarian cancer, or prostate cancer and a Dose-Expansion Phase (Part 2) in participants with advanced prostate cancer who have had at least one line of prior therapy with second-generation androgen-receptor (AR)-targeted agents (e.g., abiraterone, enzalutamide, apalutamide).

DETAILED DESCRIPTION:
There are two parts in the study. A Dose-Escalation Phase (Part 1) in participants with previously treated advanced breast cancer, ovarian cancer, or prostate cancer. There will be a 7-day run-in period with ipatasertib alone prior to Cycle 1, Day 1. After the completion of the ipatasertib run-in period, participants will begin Cycle 1, Day 1 of the ipatasertib and rucaparib combination treatment. Each cycle has 28 days. Participants will be split into 4 cohorts: Dose Level 1 group - 300 mg ipatasertib once daily (QD) + 400 mg rucaparib twice daily (BID), Dose Level 2a: 300 mg ipatasertib QD + 600 mg rucaparib BID, Dose Level 2b: 400 mg ipatasertib QD + 400 mg rucaparib BID, Dose Level 3: 400 mg ipatasertib QD + 600 mg rucaparib BID

A Dose-Expansion Phase (Part 2) - The recommended dose identified in Part 1 (highest dose level of ipatasertib and rucaparib with an acceptable safety profile and less than one-third of participants experience a dose limiting toxicity) will be evaluated in participants with advanced prostate cancer who have had at least one line of prior therapy with second-generation androgen-receptor (AR)-targeted agents (e.g., abiraterone, enzalutamide, apalutamide).

Enrollment in Cohort 3 in dose escalation phase was not opened as one-third of Dose Limiting Toxicity (DLT) evaluable participants receiving the highest dose of rucaparib in Cohort 2a experienced a DLT.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* A life expectancy of at least 3 months
* Ability to swallow oral study drug
* Have adequate organ and marrow function as confirmed by the laboratory values listed below, obtained within 28 days prior to the first dose of study treatment:
* Bone marrow function assessments (without transfusion within 28 days prior to receipt of study treatment):

  1. ANC >= 1500 cells/uL (1.5 x 10^9/L) without granulocyte-colony stimulating factor support
  2. Platelet count >= 100.0 x 10^9/L
  3. Hemoglobin >= 9 g/dL (or 5.6 mmol/L)
* Chemistry panel assessments:

  1. AST and ALT <= 1.5 x upper limit of normal (ULN); if liver metastases, <= 2.5 x ULN
  2. Bilirubin <= 1.5 x ULN (<= 3 x ULN if hyperbilirubinemia is due to Gilbert's syndrome)
  3. Serum albumin >= 3.0 g/dL
  4. Serum creatinine <= 1.5 x ULN or creatinine clearance >= 50 mL/min
  5. Fasting glucose <= 150 mg/dL and hemoglobin A1c <= 7.5%
* Resolved or stabilized toxicities resulting from previous therapy to Grade 1 (except for alopecia and neuropathy).

Cancer-Related Inclusion Criteria

* Have a histologically confirmed diagnosis of ovarian (Part 1 only), breast (Part 1 only) or prostate cancer (Part 1 and Part 2)
* Disease must be either metastatic or locally advanced disease that cannot be treated with curative intent
* For patients with ovarian cancer (Part 1 only):

  1. High-grade (2 or 3) serous or endometrioid or clear cell epithelial ovarian, fallopian tube, or primary peritoneal cancer (PPC)
  2. Must have received at least one prior platinum-based therapy and may have platinumsensitive disease (i.e., documented radiologic disease progression >= 6 months following the last dose of the platinum treatment administered) or platinum-resistant disease
  3. Have a CA-125 level that is > 2 x ULN
  4. Must have measurable disease by RECIST v1.1
* For patients with breast cancer (Part 1 only): must be human epidermal growth factor receptor 2 negative (HER2-) (estrogen receptor [ER]/progesterone positive or negative):

  1. ER/progesterone-positive patients must have received and progressed on at least one endocrine therapy (adjuvant or metastatic)
  2. ER/progesterone-negative/HER2- (triple-negative breast cancer [TNBC]) patients must have received at least one prior line of chemotherapy for metastatic breast cancer
  3. Must not have received more than two prior lines of chemotherapy for metastatic breast cancer
  4. Must have measurable disease by RECIST v1.1

For patients with prostate cancer:

1. Adenocarcinoma of the prostate without small cell or neuroendocrine features
2. Surgical or medical castration with testosterone < 50 ng/dL (1.7 nM)
3. Patients treated with luteinizing hormone-releasing hormone analogs must have initiated therapy at least 4 weeks prior to the first dose of study treatment and continue throughout the study treatment
4. Progression of prostate cancer either via PSA progression (two rising PSA levels measured >= 1 week apart, with second result >= 1 ng/mL) or radiographic progression with or without PSA progression
5. Must have received at least one prior line of second-generation androgen receptor targeted therapy (e.g., abiraterone, enzalutamide, apalutamide)
6. Patients with prostate cancer must have either measurable disease by RECIST v1.1 or bone lesions by bone scan, or both.

   * Submission of a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or a minimum of 12 freshly cut, unstained, serial tumor slides from the most recently collected tumor tissue for central molecular analysis (retrospective NGS testing for HR and PI3K-AKT pathway status and for other protocol-mandated secondary and exploratory assessments). Cytologic or fine needle aspirate samples are not acceptable. Tumor tissue from bone metastases is not acceptable.
   * For men and women of child bearing potential: agreement to remain abstinent or use protocol defined contraceptive measures during the treatment period and for at least 28 days after the last dose of ipatasertib,or 6 months after the last dose of rucaparib, whichever occurs later

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 28 days after the final dose of ipatasertib or 6 months after the final dose of rucaparib
* Prior treatment with a PARP inhibitor, AKT inhibitor, or PI3K inhibitor
* Treatment with investigational therapy within 14 days prior to initiation of study drug
* Symptomatic and/or untreated CNS metastases
* Uncontrolled tumor-related pain
* Non-study-related minor surgical procedures <= 5 days or major (invasive) surgical procedure <=14 days prior to first dose of study treatment
* Patients with active hepatitis C virus (HCV)
* Hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test or a positive quantitative HBV DNA test
* Known HIV infection
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Serious infection requiring antibiotics within 14 days of first dose of study treatment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Need for chronic corticosteroid therapy of >= 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease
* History of another malignancy within 5 years prior to randomization, except for either adequately treated non-melanomatous carcinoma of the skin, adequately treated melanoma in situ, adequately treated non-muscle-invasive urothelial carcinoma of the bladder (Tis, Ta, and low-grade T1 tumors), or other malignancies where the patient has undergone potentially curative therapy with no evidence of disease and are deemed by the treating physician to have a recurrence rate of < 5% at 5 years.
* History of clinically significant cardiovascular dysfunction
* Presence of any other condition that may have increased the risk associated with study participation or may have interfered with the interpretation of study results, and, in the opinion of the investigator, would have made the patient inappropriate for entry into the study

Ipatasertib-Specific Exclusion Criteria:

* Type 1 or Type 2 diabetes mellitus requiring insulin at study entry
* History of inflammatory bowel disease (e.g., Crohn disease and ulcerative colitis), active bowel inflammation (e.g., diverticulitis)
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 4 weeks or five elimination half-live of the inhibitors, whichever is longer, prior to initiation of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (4):
  - California Cancer Associates for Research & Excellence, Inc., San Marcos, California
  - Regional Cancer Care Associates LLC, Central Jersey Division, East Brunswick, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Medical Research Center; Oncology, Dallas, Texas
- Australia (3):
  - Kinghorn Cancer Centre; St Vincents Hospital, Darlinghurst, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Cabrini Hospital Malvern, Malvern, Victoria
- Italy (4):
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori; S. C. Oncologia Medica 2, Milan, Lombardy
  - Azienda Ospedaliera Santa Maria di Terni, Terni, Umbria
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga

REFERENCES:
- [Derived] Pook D, Geynisman DM, Carles J, de Braud F, Joshua AM, Perez-Gracia JL, Llacer Perez C, Shin SJ, Fang B, Barve M, Maruzzo M, Bracarda S, Kim M, Kerloeguen Y, Gallo JD, Maund SL, Harris A, Huang KC, Poon V, Sutaria DS, Gurney H. A Phase Ib, Open-label Study Evaluating the Safety and Efficacy of Ipatasertib plus Rucaparib in Patients with Metastatic Castration-resistant Prostate Cancer. Clin Cancer Res. 2023 Sep 1;29(17):3292-3300. doi: 10.1158/1078-0432.CCR-22-2585. PMID 37339186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in 5 countries (Australia, Italy, the Republic of Korea, Spain, and the United States) from 12 June 2019 to 04 January 2022.
Pre-assignment Details: A total of 78 participants were screened. Enrollment in Cohort 3 was not opened as one-third of Dose Limiting Toxicity (DLT) evaluable participants receiving the highest dose of rucaparib in Cohort 2a experienced a DLT.
Groups:
- Dose Escalation-Cohort 1: Participants with advanced breast cancer, ovarian cancer, or prostate cancer received ipatasertib, 300 milligrams (mg), orally, once daily (QD) for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 400 mg, orally twice daily (BID) in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2a: Participants with advanced breast cancer, ovarian cancer, or prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 600 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2b: Participants with advanced breast cancer, ovarian cancer, or prostate cancer received ipatasertib, 400 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 400 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Expansion: Participants with advanced prostate cancer received ipatasertib, 400 mg, orally QD and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator decision to withdraw, whichever occurred first.
Period: Overall Study
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Started | 8 | 6 | 7 | 30
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 7 | 30
Not completed — Death | 6 | 3 | 6 | 10
Not completed — Reason Not Specified | 2 | 2 | 1 | 15
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were treated with at least one dose of the study treatment.
Groups:
- Dose Escalation-Cohort 1: Participants with advanced breast cancer, ovarian cancer, or prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion | Total
Number analyzed (Participants) | 8 | 6 | 7 | 30 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (4.7) | 65.2 (6.0) | 69.3 (5.9) | 69.1 (9.2) | 68.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 0 | 4
  Male | 5 | 5 | 7 | 30 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Not Hispanic or Latino | 8 | 6 | 6 | 28 | 48
    Not Stated | 0 | 0 | 1 | 0 | 1
    Unknown | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian | 0 | 0 | 0 | 4 | 4
    White | 8 | 6 | 6 | 26 | 46
    Unknown | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: From Baseline up until 90 days after the last dose of study drug (up to 2 years)
Population: Safety population included all participants who were treated with at least one dose of the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 8 | 6 | 7 | 30
percentage of participants | 100 | 100 | 100 | 100

2. Primary Outcome: Dose Escalation: Percentage of Participants With Dose-Limiting Toxicities (DLTs) That Determine the Maximum-Tolerated Dose (MTD) of the Ipatasertib and Rucaparib Combination
Description: A DLT was defined as adverse events related to study treatments occurring during the DLT reporting period, which included: any death related to study treatment; grade 4 neutropenia lasting for ≥7 days; grade ≥3 neutropenia complicated by fever ≥38°C or infection; grade 4 thrombocytopenia lasting for ≥7 days; grade ≥3 thrombocytopenia complicated by hemorrhage or that requires transfusion; study treatment-related grade ≥3 non-hematologic toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5 (NCI CTCAE, v5.0).
Time Frame: Day -7 to Day 28 of Cycle 1 (1 cycle = 28 days) (up to 35 days)
Population: Safety population included all participants who were treated with at least one dose of the study treatment. Results for dose expansion is not presented.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b
Number analyzed (Participants) | 8 | 6 | 7
percentage of participants | 12.5 | 33.3 | 0

3. Primary Outcome: Percentage of Participants With Prostate-Specific Antigen Response (PSAR)
Description: PSA response was defined as the percentage of participants with a reduction in the PSA level of 50% or more. PSA response analysis was based on central PSA measurement. The 95% CI was estimated using the Clopper-Pearson method.
Time Frame: From Baseline up to 1.5 years
Population: Efficacy-evaluable population included all participants who had prostate cancer, baseline lesion, and received actual dosing equivalent to the planned dose of treatment. Number of participants analyzed are participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation-Cohort 1: Participants with advanced prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2a: Participants with advanced prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 600 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2b: Participants with advanced prostate cancer received ipatasertib, 400 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 400 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Expansion: Participants with advanced prostate cancer received ipatasertib, 400 mg, orally QD and rucaparib, 400 mg, orally BID in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or participant or investigator decision to withdraw, whichever occurred first.
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 26
percentage of participants | 0 [0.00 to 60.24] | 33.3 [0.84 to 90.57] | 25.0 [0.63 to 80.59] | 23.1 [8.97 to 43.65]

4. Secondary Outcome: Percentage of Participants With Objective Response, as Assessed by Investigator Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v.1.1)
Description: Objective response rate (ORR), defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart, as determined by the investigator per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1). A complete response was defined as the disappearance of all lesions. Pathological lymph nodes (whether target or non-target) must have a reduction in short axis to less than 10 millimeters (mm). A partial response was defined as ≥30% decrease in the sum of the diameter of target lesions, in the absence of CR persistence of one or more non-target lesions. The analysis is based on the subset of participants with measurable lesions as per RECIST criteria at baseline. ORR was calculated, and the 95% CI was estimated using the Clopper-Pearson method.
Time Frame: From Baseline up to 1.5 years (assessed at the end of Cycle 2,4,6, and every 3 cycles thereafter up to progression, 1 cycle= 28 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Expansion: Participants with advanced prostate cancer received ipatasertib, 400 mg, orally QD and rucaparib, 400 mg, orally BID 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator decision to withdraw, whichever occurred first.
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 2 | 1 | 6 | 15
percentage of participants | 0 [0.00 to 84.19] | 0 [0.00 to 97.50] | 0 [0.00 to 45.93] | 13.3 [1.66 to 40.46]

5. Secondary Outcome: Duration of Objective Response in Participants With Measurable Disease at Baseline, as Assessed by Investigator Based on RECIST v1.1
Description: DOR was defined as the time from the first occurrence of a documented objective response until the time of documented disease progression or death from any cause during the study, whichever occurred first. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and an absolute increase of at least 5 mm, or the presence of new lesions. The duration of response was estimated by Kaplan-Meier. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 4
Population: Intent-to-treat population included all participants who were treated with at least one dose of the study treatment. Number of participants analyzed is the number of participants with confirmed objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion
Number analyzed (Participants) | 2
months | NA [NA to NA] — Median upper and limit of 95% CI was not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Radiographic Progression Free Survival (rPFS), as Assessed by Prostate Cancer Working Group 3 Criteria (PCWG3)
Description: rPFS was defined as the time from study treatment initiation to the first occurrence of documented disease progression, as assessed by the investigator with the use of the PCWG3 criteria (soft tissue: Progressive disease on computed tomography [CT] or MRI scans according to RECIST v1.1, and bone metastasis by bone scan according to the PCWG3 criteria) or death from any cause, whichever occurred first. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and an absolute increase of at least 5 mm, or the presence of new lesions. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 4
Population: Efficacy-evaluable population included all participants who had prostate cancer, baseline lesion, and received actual dosing equivalent to the planned dose of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 6 | 4 | 7 | 28
months | 11.0 [9.8 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 3.0 [1.9 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 5.1 [2.1 to 11.2] | 7.2 [4.0 to 10.9]

7. Secondary Outcome: Overall Survival (OS) in All Participants
Description: OS was defined as the time from study treatment initiation to the time of death due to any cause. Kaplan-Meier method was used to estimate the median. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline to death from any cause, assessed up to 2 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Escalation-Cohort 1: Participants with prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day Cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2a: Participants with prostate cancer received ipatasertib, 300 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 300 mg, orally QD, and rucaparib, 600 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
- Dose Escalation-Cohort 2b: Participants with prostate cancer received ipatasertib, 400 mg, orally, QD for 7 days in the run-in period. Participants then received ipatasertib, 400 mg, orally QD, and rucaparib, 400 mg, orally BID in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator's decision to withdraw, whichever occurred first.
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 6 | 4 | 7 | 28
months | 20.8 [14.4 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 13.8 [4.8 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 13.3 [9.9 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [10.9 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Plasma Concentration of Ipatasertib
Time Frame: Dose Escalation: Cycle 1: Day 1 and 15 (1, 2 ,3, 5 hours post-dose), Day 15 (Predose) and Cycle 2: Day 1 and 15 (Predose); Dose Expansion: Cycle 1: Day 15 (Predose) and Cycle 2: Day 1 and 15 (Predose) (1 cycle = 28 days)
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Dose Expansion: Participants with advanced prostate cancer received ipatasertib, 400 mg, orally QD and rucaparib, 400 mg, orally BID, on Day 1, 8, and 15 in Cycle 1 in each 28-day cycle until disease progression, unacceptable toxicity, death, or participant or investigator decision to withdraw, whichever occurred first.
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 8 | 6 | 7 | 30
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1:1 hour post dose: number analyzed (Participants) | 7 | 6 | 7 | 0
  Cycle 1 Day 1:1 hour post dose | 160 (262.1) | 172 (89.2) | 192 (106.0) |
  Cycle 1 Day 1:2 hour post dose: number analyzed (Participants) | 8 | 6 | 7 | 0
  Cycle 1 Day 1:2 hour post dose | 159 (59.0) | 133 (77.7) | 230 (44.7) |
  Cycle 1 Day 1:3 hour post dose: number analyzed (Participants) | 8 | 6 | 7 | 0
  Cycle 1 Day 1:3 hour post dose | 116 (85.7) | 131 (49.0) | 249 (24.5) |
  Cycle 1 Day 1:5 hour post dose: number analyzed (Participants) | 7 | 6 | 7 | 0
  Cycle 1 Day 1:5 hour post dose | 93.4 (52.9) | 127 (58.4) | 171 (23.9) |
  Cycle 1 Day 15: Predose: number analyzed (Participants) | 7 | 4 | 6 | 25
  Cycle 1 Day 15: Predose | 21.6 (57.1) | 39.4 (178.4) | 33.5 (29.5) | 48.4 (96.6)
  Cycle 1 Day 15:1 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:1 hour post dose | 130 (126.3) | 242 (100.8) | 158 (94.8) |
  Cycle 1 Day 15:2 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:2 hour post dose | 98.7 (98.0) | 177 (119.3) | 177 (51.3) |
  Cycle 1 Day 15:3hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:3hour post dose | 92.4 (53.2) | 141 (108.7) | 181 (43.1) |
  Cycle 1 Day 15:5 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:5 hour post dose | 85.1 (28.7) | 105 (126.1) | 172 (33.1) |
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 7 | 3 | 6 | 23
  Cycle 2 Day 1: Predose | 19.2 (108.1) | 20.9 (51.3) | 40.1 (33.2) | 31.2 (226.3)
  Cycle 2 Day 15: Predose: number analyzed (Participants) | 5 | 3 | 5 | 18
  Cycle 2 Day 15: Predose | 18.9 (72.6) | 31.1 (78.0) | 49.4 (43.5) | 48.6 (77.2)

9. Secondary Outcome: Plasma Concentration of Ipatasertib's Metabolite (G-037720)
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 8 | 6 | 7 | 30
ng/mL
  Cycle 1 Day 1:1 hour post dose: number analyzed (Participants) | 7 | 6 | 7 | 0
  Cycle 1 Day 1:1 hour post dose | 65.0 (187.1) | 81.1 (81.1) | 82.0 (119.3) |
  Cycle 1 Day 1:2 hour post dose: number analyzed (Participants) | 7 | 6 | 7 | 0
  Cycle 1 Day 1:2 hour post dose | 71.2 (51.7) | 92.7 (70.6) | 115 (53.0) |
  Cycle 1 Day 1:3 hour post dose: number analyzed (Participants) | 8 | 6 | 7 | 0
  Cycle 1 Day 1:3 hour post dose | 57.8 (62.2) | 85.0 (46.2) | 141 (42.8) |
  Cycle 1 Day 1:5 hour post dose: number analyzed (Participants) | 8 | 6 | 7 | 0
  Cycle 1 Day 1:5 hour post dose | 44.0 (53.3) | 85.3 (54.3) | 112 (32.2) |
  Cycle 1 Day 15: Predose: number analyzed (Participants) | 7 | 4 | 6 | 25
  Cycle 1 Day 15: Predose | 11.8 (25.0) | 23.7 (128.8) | 20.2 (21.4) | 25.7 (103.2)
  Cycle 1 Day 15:1 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:1 hour post dose | 38.0 (111.9) | 67.4 (35.8) | 56.1 (104.8) |
  Cycle 1 Day 15:2 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:2 hour post dose | 43.2 (85.9) | 76.3 (55.4) | 65.0 (69.0) |
  Cycle 1 Day 15:3 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15:3 hour post dose | 38.5 (62.8) | 65.8 (61.9) | 75.9 (56.8) |
  Cycle 1 Day 15: 5 hour post dose: number analyzed (Participants) | 7 | 3 | 6 | 0
  Cycle 1 Day 15: 5 hour post dose | 33.0 (42.8) | 53.3 (81.9) | 73.4 (34.3) |
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 7 | 3 | 6 | 23
  Cycle 2 Day 1: Predose | 10.3 (58.0) | 13.9 (62.9) | 22.4 (35.1) | 16.3 (131.2)
  Cycle 2 Day 15: Predose: number analyzed (Participants) | 5 | 3 | 5 | 18
  Cycle 2 Day 15: Predose | 11.3 (29.9) | 19.7 (99.6) | 26.4 (38.8) | 23.6 (75.4)

10. Secondary Outcome: Plasma Concentration of Rucaparib
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1 and 15: Predose (1 cycle = 28 days)
Population: PK-evaluable population included all participants who had at least one evaluable PK sample. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
Number analyzed (Participants) | 8 | 6 | 7 | 30
ng/mL
  Cycle 1 Day 15: Predose: number analyzed (Participants) | 7 | 4 | 6 | 24
  Cycle 1 Day 15: Predose | 775 (102.3) | 3130 (142.5) | 994 (57.2) | 1660 (64.8)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 7 | 3 | 6 | 23
  Cycle 2 Day 1: Predose | 631 (178.9) | 1660 (79.1) | 1050 (57.7) | 1210 (200.1)
  Cycle 2 Day 15: Predose: number analyzed (Participants) | 6 | 5 | 5 | 21
  Cycle 2 Day 15: Predose | 1090 (51.4) | 263 (6165.7) | 1250 (48.3) | 975 (217.5)

ADVERSE EVENTS:
Time Frame: From Baseline up until 90 days after the last dose of study drug (up to 2 years)
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Dose Escalation-Cohort 1 | Dose Escalation-Cohort 2a | Dose Escalation-Cohort 2b | Dose Expansion
All-Cause Mortality (participants affected / at risk) | 6/8 | 3/6 | 6/7 | 10/30
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 1/7 | 8/30
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 7/7 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation-Cohort 1 (N=8) | Dose Escalation-Cohort 2a (N=6) | Dose Escalation-Cohort 2b (N=7) | Dose Expansion (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation-Cohort 1 (N=8) | Dose Escalation-Cohort 2a (N=6) | Dose Escalation-Cohort 2b (N=7) | Dose Expansion (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (6) | 1 (1) | 9 (12)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 7 (16) | 6 (13) | 6 (14) | 29 (65)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 5 (12) | 5 (9) | 20 (35)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (6) | 4 (4) | 11 (15)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 9 (10)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (5) | 4 (7) | 3 (5) | 17 (19)
Hernia pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (5) | 1 (2) | 10 (13)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 7 (12)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 3 (4)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 4 (6)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 3 (3) | 5 (5) | 2 (3) | 18 (18)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 3 (5) | 1 (1) | 16 (21)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03840200/Prot_SAP_000.pdf